CLINICAL TRIAL: NCT02463409
Title: Effects of Theophylline on cAMP Signaling in Children With Pseudohypoparathyroidism Type 1a
Brief Title: Theophylline as a Treatment for Children With Pseudohypoparathyroidism Type 1a (Albright Hereditary Osteodystrophy)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ashley Shoemaker, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 150497
Record Dates: First submitted 2015-05-20; First posted 2015-06-04 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Pseudohypoparathyroidism Type 1a; Albright Hereditary Osteodystrophy
MeSH Terms: conditions — Pseudohypoparathyroidism | interventions — Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Theophylline (Experimental): Patients will receive a 24 hour continuous infusion of intravenous theophylline.
  Interventions: Drug: Theophylline

INTERVENTIONS:
Drug: Theophylline — 24 hour infusion of IV theophylline
  Other Names: Theo

SUMMARY:
This study will test an investigational drug, theophylline, in children with pseudohypoparathyroidism type 1a (PHP1a). This study involves a 3 day visit to the Vanderbilt Clinical Research Center.

DETAILED DESCRIPTION:
Study measures will be done at baseline and during a 24h infusion of IV theophylline. Theophylline levels will be drawn to ensure therapeutic dosing and to monitor for toxicity. Measures include laboratory values, response to PTH infusion and resting energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10 to 21 years old
2. English proficiency
3. Clinical and genetic diagnosis of PHP1a

Exclusion Criteria:

1. Use of a PDE inhibitor in the past 30 days
2. History of a seizure disorder unrelated to hypocalcemia
3. History of a cardiac arrhythmia (not including bradycardia)
4. History of hepatic insufficiency
5. AST or ALT >2x upper limit of normal
6. Total bilirubin >1.5 x upper limit of normal (unless patient has a diagnosis of Gilbert's syndrome and no other causes leading to hyperbilirubinemia are identified)
7. Congestive heart failure
8. Cigarette use in the past 30 days
9. Alcohol use within the past 24 hours
10. Current pregnancy
11. Untreated hypothyroidism (defined as free T4 level < 0.6 ng/dL or TSH >10 mcU/mL)
12. Active peptic ulcer disease
13. Fever >101 degrees in the past 24 hours
14. Current use of medications known to effect theophylline levels (listed below)
15. Severe sleep apnea requiring BiPAP

Drugs with clinically significant drug interactions with theophylline:

* Allopurinol
* Cimetidine
* Ciprofloxacin
* Clarithromycin
* Enoxacin
* Ephedrine
* Erythromycin
* Estrogen
* Flurazepam
* Fluvoxamine
* Lithium
* Lorazepam
* Methotrexate
* Midazolam
* Pentoxifylline
* Propranolol
* Rifampin
* Sulfinpyrazone
* Tacrine
* Thiabendazole
* Ticlopidine
* Troleandomycin
* Verapamil

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley H Shoemaker, MD, MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Unversity, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators may contact Dr. Shoemaker for data after our primary analysis is completed and published (if applicable).

REFERENCES:
- [Background] Landreth H, Malow BA, Shoemaker AH. Increased Prevalence of Sleep Apnea in Children with Pseudohypoparathyroidism Type 1a. Horm Res Paediatr. 2015;84(1):1-5. doi: 10.1159/000381452. Epub 2015 Apr 23. PMID 25925491
- [Background] Shoemaker AH, Lomenick JP, Saville BR, Wang W, Buchowski MS, Cone RD. Energy expenditure in obese children with pseudohypoparathyroidism type 1a. Int J Obes (Lond). 2013 Aug;37(8):1147-53. doi: 10.1038/ijo.2012.200. Epub 2012 Dec 11. PMID 23229731
- See also: Vanderbilt PHP Research Page — http://www.facebook.com/pseudohypoparathyroidism

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The screening visit included labs, physical exam and medical history, prior to assignment to the theophylline arm.
Period: Overall Study
Arm/Group | Theophylline
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Population: All patients who enrolled in the study, not including screen fails
Arm/Group | Theophylline
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Urine cAMP
Description: Change in urine cAMP (after parathyroid hormone stimulation) before and during treatment with theophylline
Time Frame: 1 day
Population: Patients treated with theophylline who maintained appropriate IV access. Only 3 patients had complete data available.
Measure: Mean (Standard Deviation); unit: fm/uL
Arm/Group | Theophylline
Number analyzed (Participants) | 3
fm/uL | 3048 (8369)

2. Secondary Outcome: Change in Resting Energy Expenditure (REE)
Description: Change in REE before and during treatment with theophylline
Time Frame: 1 day
Measure: Mean (Standard Error); unit: kcals per day
Arm/Group | Theophylline
Number analyzed (Participants) | 4
kcals per day | -14 (68)

3. Secondary Outcome: Change in Apnea Hypopnea Index (AHI)
Description: Change in AHI before and during treatment with theophylline
Time Frame: 1 day
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Theophylline
Number analyzed (Participants) | 4
units on a scale | -0.60 (0.67)

ADVERSE EVENTS:
Time Frame: 3 days
Description: We specifically asked patients about headache, nausea and vomiting at least twice daily. They were monitored continuously via telemetry for arrhythmia. Other adverse events were reported as described by the partiicipant.
Groups:
- Theophylline: Patients will receive a 24 hour continuous infusion of intravenous theophylline.
  Theophylline: 24 hour infusion of IV theophylline. All patients who enrolled in the study are included in this group (excluding screen fails).
Arm/Group | Theophylline
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theophylline (N=5)
Nausea (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes